CLINICAL TRIAL: NCT00920738
Title: Metabolic Syndrome in Childhood Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2003NT064; 0411M65666 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Brain and Central Nervous System Tumors; Leukemia; Lymphoma; Metabolic Syndrome; Sarcoma
Keywords: metabolic syndrome; cancer survivor; childhood soft tissue sarcoma; unspecified childhood solid tumor, protocol specific; childhood acute lymphoblastic leukemia; childhood chronic myelogenous leukemia; childhood Hodgkin lymphoma; childhood non-Hodgkin lymphoma; childhood acute myeloid leukemia/other myeloid malignancies; chronic lymphocytic leukemia; childhood brain stem glioma; childhood cerebellar astrocytoma; childhood cerebral astrocytoma/malignant glioma; childhood choroid plexus tumor; childhood craniopharyngioma; childhood embryonal tumor; childhood ependymoma; childhood oligodendroglioma; childhood pineal parenchymal tumor; childhood mixed glioma; childhood subependymal giant cell astrocytoma; childhood visual pathway and hypothalamic glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Lymphoma; Metabolic Syndrome; Sarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Astrocytoma; Choroid Plexus Neoplasms; Familial ependymoma; Oligodendroglioma; Optic Nerve Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 22 gauge intravenous polyethylene catheter will be inserted into an antecubital vein of one arm and the necessary blood for all baseline laboratory studies will be obtained and processed as per standard protocol.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cancer Survivors: Subjects who are cancer survivors must have survived childhood cancer (diagnosed < or = 18 years) for a minimum of 5 years and be in remission.
  Interventions: Other: metabolic assessment; Other: questionnaire administration
- Healthy Siblings of Cancer Survivor: Healthy populations similar in age and gender distribution, derived from a frequency matched control population of 350 healthy siblings.
  Interventions: Other: metabolic assessment; Other: questionnaire administration

INTERVENTIONS:
Other: metabolic assessment — Physical examination, medical history, blood pressure, anthropometrics, laboratory studies and other procedures (body composition, bone density, growth hormone, vascular, functional mobility, body fat assessments, etc).
Other: questionnaire administration — Dietary habits will be evaluated using the Youth/ Adolescent Questionnaire (YAQ)and the Modifiable Activity Questionnaire for Adolescents (MAQA) will be used to assess participation in leisure time and competitive activities during the past year will be administered on Day 2.
  Other Names: MAQA; AQA

SUMMARY:
RATIONALE: Gathering information about how often metabolic syndrome occurs in young survivors of childhood cancer may help doctors learn more about the disease.

PURPOSE: This clinical trial is studying metabolic syndrome in survivors of childhood cancer and in their healthy sisters and brothers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the manifestations of metabolic syndrome (MS) in children and adolescents who are survivors of childhood cancer (CCS).
* Compare the prevalence of MS in CCS to that of matched healthy siblings of similar age and gender.
* Evaluate insulin resistance (as measured by the euglycemic insulin clamp) in CCS and compare to that of healthy siblings of similar age and gender.
* Assess the extent to which prevalent obesity and insulin resistance are correlated with other factors that have been identified in the causal pathway associated with the development of the MS that may be altered in the CCS ( e.g., growth-hormone secretion, adipokines [adiponectin, leptin], inflammatory mediators [e.g., interleukin-6], tumor necrosis factor-α, and C-reactive protein).
* Obtain dietary and physical activity assessments of CCS and healthy siblings.

Secondary

* Explore demographic (age at treatment, sex-specific differences) and treatment-related factors (exposures and dose-related associations with chemotherapeutic agents, radiation, steroids) as potential correlates with insulin resistance, vascular function, and MS in CCS.

OUTLINE: Patients undergo a comprehensive medical examination including current and past medical history, family history, review of prescription medications, a physical examination including a body and visceral-fat assessment, and anthropometric (DEXA and bone-age x-ray) and blood pressure measurement. Blood samples are collected to measure growth hormone, adipokines (adiponectin, leptin), cytokines (IL-6 and CRP), fasting insulin, fasting glucose, lipids, oxidized LDL, hypothalami-pituitary-gonadal function (estrogen, FSH, LH, testosterone), and thyroid function (free T4 and TSH). Patients also complete questionnaires on dietary intake and physical activity.

Healthy siblings undergo a complete medical examination as patients do, including blood samples collection and questionnaire administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be survivors of childhood cancer, treated at Fairview-University Medical Center or Children's Hospitals and Clinics of Minneapolis and St Paul or siblings of survivors.
* Subjects will be 9-17 years old at the time of their visit.
* Subjects who are cancer survivors must have survived childhood cancer for a minimum of 5 years and be in remission.

Exclusion Criteria:

* Eligibility will not be restricted by race or sex.
* Any women currently pregnant will not be eligible, but may participate 3 or more months after the end of her pregnancy if the study is still ongoing.
* Subjects who underwent hematopoietic cell transplant (HCT) are not eligible for this study.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The childhood cancer survivor (CCS) subjects for this study will be selected from Pediatric Oncology databases at the University of Minnesota Medical Center and Children"s Hospitals and Clinics of Minneapolis and St. Paul as described previously. CCS will complete a comprehensive evaluation in the Masonic Clinical Research Unit (MCRU) over a 2 day time period. The comparative data on normal children and adolescents will be obtained from healthy siblings frequency matched by age and gender and who will be evaluated in a manner similar to the CCS.
Sampling Method: Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2005-04; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome (MS) in survivors of childhood cancer (CCS) vs controls | Day 1 and Day 2
Insulin resistance (IR) in CCS vs controls | Day 1 and Day 2
Correlation of obesity and IR to other factors associated with the development of the MS that may be altered in the CCS | Day 1 and Day 2
Dietary and a physical activity assessments of CCS vs controls | Day 1 and Day 2

SECONDARY OUTCOMES:
Demographic and treatment-related factors as potential correlates with IR, vascular function, and MS in CCS | Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Julia Steinberger, MD, MS, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Children's Hospital - Fairview, Minneapolis, Minnesota, United States